CLINICAL TRIAL: NCT05820633
Title: Pelvic Nodes Ultra-Hypo Fractionated Versus Conventionally Fractionated IMRT With HDR Brachytherapy Boost in Prostate Cancer: A Collaborative Multi-institutional Non-inferiority Phase 3 Trial. (PCS-XI)
Brief Title: Pelvic Nodes Ultra-Hypo vs Conventionally Fractionated IMRT With HDR Boost in Prostate Cancer.
Acronym: PCS-XI
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: amendment to be done, adding 200 patients
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: TerSera Therapeutics LLC (Industry)
Responsible Party: Principal Investigator, André-Guy Martin, Principal Investigator, M.D., M.Sc., F.R.C.P.C., CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-20-2023-6396: PCS XI
Record Dates: First submitted 2023-02-26; First posted 2023-04-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Node; Prostate; Radiotherapy Side Effect
Keywords: ultra hypo fractionation; brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Menogaril

STUDY DESIGN:
Intervention Model Description: randomized phase 3 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultra hypo fractionation radiation therapy (UHF) (Experimental): 5 radiation treatments (5 Gy per fraction) to the prostate, seminal vesicle and pelvic nodes given every other day over 2 weeks for a total of 25 Gy.
  Interventions: Radiation: Report and compare changes in a non-inferiority analysis of the International Prostate Symptom Score (I-PSS); Radiation: Report and compare changes in a non-inferiority analysis of the expanded prostate cancer index composite" (EPIC-26):; Radiation: Report and compare changes in a non-inferiority analysis of the Sexual Health Inventory for Men (SHIM); Radiation: Report and compare changes in a non-inferiority analysis of the toxicities reported according to the Common Terminology Criteria for Adverse Events (CTCAE); Radiation: Report and compare the biochemical disease free survival (bDFS); Radiation: Report and compare the disease free survival (DFS); Radiation: Report and compare the metastase free survival (MFS); Radiation: Report and compare the overall survival (OS)
- standard of care fractionation (SOC) (Active Comparator): 20-25 radiation treatments (range: 1,8 to 2,15 Gy per fraction) to the prostate, seminal vesicle and pelvic nodes given in 20-25 working day treatments over 4-5 weeks for a total of 43 Gy to 46 Gy.
  Interventions: Radiation: Report and compare changes in a non-inferiority analysis of the International Prostate Symptom Score (I-PSS); Radiation: Report and compare changes in a non-inferiority analysis of the expanded prostate cancer index composite" (EPIC-26):; Radiation: Report and compare changes in a non-inferiority analysis of the Sexual Health Inventory for Men (SHIM); Radiation: Report and compare changes in a non-inferiority analysis of the toxicities reported according to the Common Terminology Criteria for Adverse Events (CTCAE); Radiation: Report and compare the biochemical disease free survival (bDFS); Radiation: Report and compare the disease free survival (DFS); Radiation: Report and compare the metastase free survival (MFS); Radiation: Report and compare the overall survival (OS)

INTERVENTIONS:
Radiation: Report and compare changes in a non-inferiority analysis of the International Prostate Symptom Score (I-PSS) — Assess early and late genito-urinary (GU) toxicities induced assessed via the International Prostate Symptom Score (I-PSS) in the experimental UHF group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group).
Radiation: Report and compare changes in a non-inferiority analysis of the expanded prostate cancer index composite" (EPIC-26): — Assess early and late genito-urinary (GU) and gastro-intestinal (GI) toxicities induced and quality of life assessed via expanded prostate cancer index composite (EPIC-26) in the experimental UHF group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group).
Radiation: Report and compare changes in a non-inferiority analysis of the Sexual Health Inventory for Men (SHIM) — Assess early and late sexual health in the experimental UHF group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group).
Radiation: Report and compare changes in a non-inferiority analysis of the toxicities reported according to the Common Terminology Criteria for Adverse Events (CTCAE) — Assess early and late toxicities reported according to the Common Terminology Criteria for Adverse Events (CTCAE) in the experimental UHF group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group).
Radiation: Report and compare the biochemical disease free survival (bDFS) — Assess the 5 and 10 years biochemical disease-free survival (bDFS) in the UHF group and compare them for non-inferiority to those of the control group.
Radiation: Report and compare the disease free survival (DFS) — Assess the 5 and 10 years disease-free survival (DFS) in the UHF group and compare them for non-inferiority to those of the control group.
Radiation: Report and compare the metastase free survival (MFS) — Assess the 5 and 10 years metastasis-free survival (MFS) in the UHF group and compare them for non-inferiority to those of the control group.
Radiation: Report and compare the overall survival (OS) — Assess the 5 and 10 years overall survival (OS) in the UHF group and compare them for non-inferiority to those of the control group.

SUMMARY:
Randomized Phase III study, comparing pelvic ultra-hypo fractionated radiotherapy (UHF: 5Gy/fraction) to a standard or moderate hypo-fractionation (1.8-2.15Gy/fraction), both associated to an HDR prostate +/- adjacent seminal vesicles brachytherapy boost (HDR-BT)+ ADT according to NCCN guidelines. Considering that the calculated bio-equivalent doses to the tumor are similar for all treatment options, the UHF technique is deemed to be non-inferior to the standard approach. Treatment acceptability, tolerance and adverse events will be reported and compared for non-inferiority as the primary objective. Secondary objectives are biochemical control, metastasis-free, disease specific and overall survival.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-skin cancer in North American men. In 2020, an estimated 23 300 Canadian men will be diagnosed with prostate cancer of which, 4200 will die. Fortunately, with an early screening, most will have a localized disease at diagnosis. Despite this, high risk disease affects a growing portion of the population and this according to age (29.3%, 39.1%, 60.4%, et 90.6% respectively at 55-59, 65-69, 75-79, & 85-89 years of age). Gleason score 8 to 10 tumors follow the same pattern (16.5%, 23.4%, 37.2%, and 59.9% at respective ages). Those patients are at risk for harboring lymph nodes metastasis.

Multiple therapeutic options, with similar biochemical disease-free survival (bDFS) are available: surgery +/- salvage radiotherapy +/- androgen deprivation therapy (ADT) or radiotherapy (RT) +/- HDR-BT +/- ADT. For men with high-risk disease, the combined approach of RT + HDR-BT + ADT might even offer higher cancer specific survival (CSS) rates when compared to surgery.

HDR-BT allows for the delivery of a very high (ablative) dose of radiation while giving a lower dose to the nearby organs at risk (OARs). Recently published literature showed that pelvic RT plus HDR-BT significantly increased bDFS (84 vs 77%).

Pelvic RT is generally given on a daily basis (5 days/week) over a period of 4-5 weeks, with 1,8-2,15Gy per fraction. This requires a substantial time investment from patients undergoing treatment. Many studies have shown that prostate cancer offers a radiation cell kill ratio (α/β) of 0.9-1.5 Gy. Furthermore, the most commonly used α/β value for prostate cancer is 1,5 Gy (range 0,8 - 2,2). This low α/β ratio offers a more efficient cell kill with hypo-fractionated doses, offering a better tumor control with a lower cumulative dose, given in a shorter time span. Recently, a multicentric randomized phase III study has shown similar late toxicity and oncologic control outcomes between UHF (>/= 5 Gy/fraction) and conventionally fractionated RT. However, until now, no phase III study has compared combined UHF pelvic RT to standard fractionation combined with an HDR-BT in this population.

The proposed experimental fractionation scheme for whole pelvic RT in this study will be 5Gy administered every other day over 2 weeks (UHF). It will be compared to standard pelvic RT (1.8-2.15Gy/working day) given over 4 to 5 weeks. Both will be combined with a single 15 Gy fraction of HDR-BT and ADT (goserelin). The UHF treatment modality significantly reduces the overall treatment time, freeing machine-time and allowing more patients to be treated. Given its low α/β ratio, prostate cancer is readily amenable to UHF fractionation. The bio-equivalent dose calculations were done based on published litterature. Neo-adjuvant and adjuvant ADT (goserelin) will be administered for a duration according to NCCN guidelines.

In these COVID-19 pandemic times, a reduction in the number of patients' visits to the clinic is highly desirable in order to limit the risk of virus transmission. UHF would also lower the socio-economic burden incurred by the patients and their families. It also increases the therapeutic efficiency reducing costs for both, patients and health services. The proposed study aims to demonstrate the non-inferiority of UHF treatment compared to standard of care. If this hypothesis is confirmed, all future patients could benefit from it.

In order to improve the quality of life of men diagnosed with prostate cancer this study aim to demonstrate that combined UHF pelvic RT plus HDR-BT (+ ADT according to NCCN guidelines) is safe and non-inferior to standard fractionation regimens in regard to toxicities and tumor control for prostate cancer patients with risk of nodal involvement. Therefore, 500 men will be recruited, in order to confirm the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed adenocarcinoma of the prostate.
* All clinical stages with lymph node involvement risk needing pelvis RT.
* Stage Mx or M0.
* Unfavorable Intermediate, high or very high-risk disease according to NCCN guidelines.
* Having the ability to give free and informed consent.

Exclusion Criteria:

* Clinical stage M1.
* IPSS Score > 20 with alpha-blocking medication.
* Prior pelvic radiotherapy,
* History of active collagenosis (Lupus, Scleroderma, Dermatomyositis).
* Past history of Inflammatory Bowell Disease.
* Bilateral hip prosthesis.

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority analysis of early change in genito-urinary (GU) toxicities induced. | Every 3 months for 1 year.
  Assess early genito-urinary (GU) toxicities induced opposed to baseline assessed via the International Prostate Symptom Score (I-PSS) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group).
Non-inferiority analysis of early change in reported Expanded Prostate Cancer Index Composite (EPIC-26) questionnaire. | Every 3 months for 1 year.
  Assess early health-related quality of life opposed to baseline assessed via the Expanded Prostate Cancer Index Composite (EPIC-26) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group) every 3 months for 1 year.
Non-inferiority analysis of late change in genito-urinary (GU) toxicities induced. | Every 6 months up to 36 months, then annually up to 10 years.
  Assess late genito-urinary (GU) toxicities induced opposed to baseline evaluated by the International Prostate Symptom Score (I-PSS) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group).
Non-inferiority analysis of late change in reported Expanded Prostate Cancer Index Composite (EPIC-26) questionnaire. | Every 6 months up to 36 months, then annually up to 10 years.
  Assess late health-related quality of life opposed to baseline assessed via the Expanded Prostate Cancer Index Composite (EPIC-26) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group) every 6 months up to 36 months, then annually.
Non-inferiority analysis of early change in sexual health. | Every 3 months for 1 year.
  Assess early quality of life opposed to baseline assessed via the Sexual Health Inventory for Men (SHIM) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group) every 3 months for 1 year.
Non-inferiority analysis of late change in sexual health. | Every 6 months up to 36 months, then annually up to 10 years.
  Assess early sexual health status opposed to baseline assessed via the Sexual Health Inventory for Men (SHIM) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group) every 6 months up to 36 months, then annually.
Non-inferiority analysis of early change in toxicities reporte via the Common Terminology Criteria for Adverse Events (CTCAE). | Every 3 months for 1 year.
  Assess early reported toxicities opposed to baseline assessed via the Common Terminology Criteria for Adverse Events (CTCAE) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group) every 3 months for 1 year, every 6 months up to 36 months, then annually.
Non-inferiority analysis of late change in toxicities reporte via the Common Terminology Criteria for Adverse Events (CTCAE). | Every 6 months up to 36 months, then annually up to 10 years.
  Assess early reported toxicities opposed to baseline assessed via the Common Terminology Criteria for Adverse Events (CTCAE) in the experimental UH group has compared in a non-inferiority analysis to those of patients who received a standard treatment (control group) every 3 months for 1 year, every 6 months up to 36 months, then annually.

SECONDARY OUTCOMES:
Non-inferiority analysis of 5 years biochemical Disease Free Survival. | 5 years (median)
  Assess the 5 years the biochemical disease-free survival (bDFS) in the UH group and compare them for non-inferiority to those of the control group.
Non-inferiority analysis of 5 years Disease Free Survival. | 5 years (median)
  Assess the 5 years the disease-free survival (DFS) in the UH group and compare them for non-inferiority to those of the control group.
Non-inferiority analysis of 5 years Metastasis Free Survival. | 5 years (median)
  Assess the 5 years the Metastasis Free Survival (MFS) in the UH group and compare them for non-inferiority to those of the control group.
Non-inferiority analysis of 5 years Overall Survival. | 5 years (median)
  Assess the 5 years the Overall Survival (OS) in the UH group and compare them for non-inferiority to those of the control group.
Non-inferiority analysis of 10 years biochemical Disease Free Survival. | 10 years (median)
  Assess the 10 years the biochemical disease-free survival (bDFS) in the UH group and compare them for non-inferiority to those of the control group.
Non-inferiority analysis of 10 years Disease Free Survival. | 10 years (median)
  Assess the 10 years the disease-free survival (DFS) in the UH group and compare them for non-inferiority to those of the control group.
Non-inferiority analysis of 10 years Metastasis Free Survival. | 10 years (median)
  Assess the 10 years the Metastasis Free Survival (MFS) in the UH group and compare them for non-inferiority to those of the control group.
Non-inferiority analysis of 10 years Overall Survival. | 10 years (median)
  Assess the 10 years the Overall Survival (OS) in the UH group and compare them for non-inferiority to those of the control group.

OTHER OUTCOMES:
Seric Testosterone change. | From baseline (randomisation), then every 3 months for 3 years, every 6 months for 2 years, and annually up to 10 years.
  Testosterone blood level, every 3 months for 3 years, every 6 months for 2 years, then annually.
Complete blood count. | Baseline prior treatment.
  Complete blood count.
Alkaline Phosphatase. | Baseline prior treatment.
  Alkaline Phosphatase blood level.
Blood urea nitrogen (BUN) | Baseline prior treatment.
  Serum creatinine to evaluate renal function.
Serum creatinine | Baseline prior treatment.
  Serum creatinine to evaluate renal function.
Concomitant added medications list. | Every 3 months for 3 years, every 6 months for 2 years, then annually up to 10 years.
  List of added medications (name and dosage) needed to alleviate symptoms of potential side effects of therapy and evolution of disease.
Treatment related loss of income evaluation in dollars estimated through the economic questionnaire. | Baseline and Month 3.
  Evaluate loss of outcomes (dollars) due to treatment
Total body bone scan in order to evaluate if bony metastasis are present or not. | Baseline prior treatment.
  Tumor extension description if presence of bony metastasis or not (for staging purposes)
Abdomino-Pelvis (thorax not compulsory) CT Scan in order to evaluate if metastasis are present or not. | Baseline prior treatment.
  Abdominal + Pelvis (thorax not compulsory) for tumor extension description =determination if presence of distant metastasis or not (for staging purposes)
Osteodensitometry. | Baseline within the first year.
  Bone density evaluation to prevent osteoporosis
Prostate MRI scan in order to evaluate if extra capsular tumor extension are present or not. | Baseline prior treatment.
  Recommended but not compulsory - Prostate MRI (tumor description of dominant involved lesion) for determination if presence extension extra capsulary or not.
Total body PET scan in order to evaluate if metastasis are present or not. | Baseline prior treatment.
  Optional (tumor extension description if presence of metastasis or not)

CONTACTS AND LOCATIONS:
Overall Officials: Andre-Guy Martin, MD MSc FRCPC, Principal Investigator — Andre-Guy Martin MD Inc.
Locations (11):
- Canada (11):
  - BC Cancer Sindi Ahluwalia centre for the Southern Interior, Kelowna, British Columbia
  - Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Lakeridge Health Oshawa Cancer centre, Oshawa, Ontario
  - CISSS de l'Outaouais, Hôpital de Gatineau, Gatineau, Quebec
  - CISSS de Laval, Hôpital de la Cité-de-la-Santé, Laval, Quebec
  - CISSS de la Montérégie-Centre, Hôpital Charles-Le Moyne, Longueuil, Quebec
  - CIUSSS du Centre-Ouest-de-l'Île-de-Montréal, Jewish General Hospital, Montreal, Quebec
  - Cedars Cancer Centre, McGill University Health Centre (MUHC), Montreal, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Hôpital Maisonneuve-Rosemont, Montreal East, Quebec
  - CIUSSS de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - CHU de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huynh-Le MP, Myklebust TA, Feng CH, Karunamuni R, Johannesen TB, Dale AM, Andreassen OA, Seibert TM. Age dependence of modern clinical risk groups for localized prostate cancer-A population-based study. Cancer. 2020 Apr 15;126(8):1691-1699. doi: 10.1002/cncr.32702. Epub 2020 Jan 3. PMID 31899813
- [Background] Heidenreich A, Varga Z, Von Knobloch R. Extended pelvic lymphadenectomy in patients undergoing radical prostatectomy: high incidence of lymph node metastasis. J Urol. 2002 Apr;167(4):1681-6. PMID 11912387
- [Background] Greenberger BA, Zaorsky NG, Den RB. Comparison of Radical Prostatectomy Versus Radiation and Androgen Deprivation Therapy Strategies as Primary Treatment for High-risk Localized Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol Focus. 2020 Mar 15;6(2):404-418. doi: 10.1016/j.euf.2019.11.007. Epub 2019 Dec 5. PMID 31813810
- [Background] Yin M, Zhao J, Monk P, Martin D, Folefac E, Joshi M, Jin N, Mortazavi A, Verschraegen C, Clinton S. Comparative effectiveness of surgery versus external beam radiation with/without brachytherapy in high-risk localized prostate cancer. Cancer Med. 2020 Jan;9(1):27-34. doi: 10.1002/cam4.2605. Epub 2019 Nov 7. PMID 31697452
- [Background] Tharmalingam H, Tsang Y, Choudhury A, Alonzi R, Wylie J, Ahmed I, Henry A, Heath C, Hoskin PJ. External Beam Radiation Therapy (EBRT) and High-Dose-Rate (HDR) Brachytherapy for Intermediate and High-Risk Prostate Cancer: The Impact of EBRT Volume. Int J Radiat Oncol Biol Phys. 2020 Mar 1;106(3):525-533. doi: 10.1016/j.ijrobp.2019.09.044. Epub 2019 Oct 11. PMID 31610249
- [Background] Morton G, Loblaw A, Cheung P, Szumacher E, Chahal M, Danjoux C, Chung HT, Deabreu A, Mamedov A, Zhang L, Sankreacha R, Vigneault E, Springer C. Is single fraction 15 Gy the preferred high dose-rate brachytherapy boost dose for prostate cancer? Radiother Oncol. 2011 Sep;100(3):463-7. doi: 10.1016/j.radonc.2011.08.022. Epub 2011 Sep 14. PMID 21924511
- [Background] Hill RP, Rodemann HP, Hendry JH, Roberts SA, Anscher MS. Normal tissue radiobiology: from the laboratory to the clinic. Int J Radiat Oncol Biol Phys. 2001 Feb 1;49(2):353-65. doi: 10.1016/s0360-3016(00)01484-x. PMID 11173128
- [Background] Williams MV, Denekamp J, Fowler JF. A review of alpha/beta ratios for experimental tumors: implications for clinical studies of altered fractionation. Int J Radiat Oncol Biol Phys. 1985 Jan;11(1):87-96. doi: 10.1016/0360-3016(85)90366-9. PMID 3881377
- [Background] McCammon R, Rusthoven KE, Kavanagh B, Newell S, Newman F, Raben D. Toxicity assessment of pelvic intensity-modulated radiotherapy with hypofractionated simultaneous integrated boost to prostate for intermediate- and high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2009 Oct 1;75(2):413-20. doi: 10.1016/j.ijrobp.2008.10.050. Epub 2009 Apr 11. PMID 19362783
- [Background] Widmark A, Gunnlaugsson A, Beckman L, Thellenberg-Karlsson C, Hoyer M, Lagerlund M, Kindblom J, Ginman C, Johansson B, Bjornlinger K, Seke M, Agrup M, Fransson P, Tavelin B, Norman D, Zackrisson B, Anderson H, Kjellen E, Franzen L, Nilsson P. Ultra-hypofractionated versus conventionally fractionated radiotherapy for prostate cancer: 5-year outcomes of the HYPO-RT-PC randomised, non-inferiority, phase 3 trial. Lancet. 2019 Aug 3;394(10196):385-395. doi: 10.1016/S0140-6736(19)31131-6. Epub 2019 Jun 18. PMID 31227373
- [Background] Arcangeli G, Saracino B, Gomellini S, Petrongari MG, Arcangeli S, Sentinelli S, Marzi S, Landoni V, Fowler J, Strigari L. A prospective phase III randomized trial of hypofractionation versus conventional fractionation in patients with high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Sep 1;78(1):11-8. doi: 10.1016/j.ijrobp.2009.07.1691. Epub 2010 Jan 4. PMID 20047800
- [Background] D'Amico AV, Chen MH, Renshaw AA, Loffredo M, Kantoff PW. Androgen suppression and radiation vs radiation alone for prostate cancer: a randomized trial. JAMA. 2008 Jan 23;299(3):289-95. doi: 10.1001/jama.299.3.289. PMID 18212313
- [Background] Partin AW, Mangold LA, Lamm DM, Walsh PC, Epstein JI, Pearson JD. Contemporary update of prostate cancer staging nomograms (Partin Tables) for the new millennium. Urology. 2001 Dec;58(6):843-8. doi: 10.1016/s0090-4295(01)01441-8. PMID 11744442
- [Background] Hall WA, Paulson E, Davis BJ, Spratt DE, Morgan TM, Dearnaley D, Tree AC, Efstathiou JA, Harisinghani M, Jani AB, Buyyounouski MK, Pisansky TM, Tran PT, Karnes RJ, Chen RC, Cury FL, Michalski JM, Rosenthal SA, Koontz BF, Wong AC, Nguyen PL, Hope TA, Feng F, Sandler HM, Lawton CAF. NRG Oncology Updated International Consensus Atlas on Pelvic Lymph Node Volumes for Intact and Postoperative Prostate Cancer. Int J Radiat Oncol Biol Phys. 2021 Jan 1;109(1):174-185. doi: 10.1016/j.ijrobp.2020.08.034. Epub 2020 Aug 27. PMID 32861817
- [Background] Gregoire JP, Moisan J, Labrecque M, Cusan L, Diamond P. [Validation of a French adaptation of the international prostatic symptom score]. Prog Urol. 1996 Apr;6(2):240-9. French. PMID 8777417
- See also: Canadian Cancer Society, statistics on prostate cancer — https://www.cancer.ca/fr-ca/cancer-information/cancer-type/prostate/statistics
- Available data/document: Study Protocol — https://www.sealedenvelope.com/simple-randomiser/v1/lists